CLINICAL TRIAL: NCT03032666
Title: Sofosbuvir/Ledipasvir for Hepatitis C Genotype 1-6 in Patients With Transfusion-Dependent Thalassemia: An Open Label Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ala'a Sharara (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Ala'a Sharara, Professor, Head of Gastroenterology Department, American University of Beirut Medical Center
Organization: American University of Beirut Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM.AS1.47
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Thalassemia; Hepatitis C
Keywords: Thalassemia; HCV; Sofosbuvir; Ledipasvir
MeSH Terms: conditions — Thalassemia; Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- sofosbuvir/velpatasvir (Experimental): Epclusa
  Interventions: Drug: sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir — treatment of hepatitis C genotype 1-6 in patients with transfusion-dependent thalassemia.
  Other Names: Epclusa

SUMMARY:
Sustained Viral Response following 12-week therapy (SVR 12) with sofosbuvir/ledipasvir in transfusion-dependent patients with HCV genotype 1-6

Secondary Objective(s):

Assessment of transfusion requirements Adverse events Efficacy in treatment-naïve vs. relapsers vs. null responders Efficacy in patients with advanced fibrosis/cirrhosis vs. F1, F2 by elastography

DETAILED DESCRIPTION:
Thalassemia is characterized by a defect in red blood cell production. The anemia is caused by destruction of the erythroblasts in the bone marrow, erythrocytes' hemolysis and disrupted erythropoiesis. The life-long need for transfusions makes patients vulnerable to transfusion transmitted viral infections especially hepatitis C virus (HCV). HCV infection is a widespread disease. It affects a large number of thalassemia patients and it is considered a major public health problem. Infection with HCV results in chronic infection in a huge proportion of infected individuals. Therefore, it has been suggested that early treatment of acute HCV may prevent the development of chronic hepatitis.

Several studies have dwelled on the efficacy of interferon therapy for acute HCV infection in adults. Newer pegylated interferons (PEG-IFN) were used in the treatment of adults with acute HCV which showed equally excellent results. However, in thalassemia patients, iron overload in the liver negatively affects the outcome of liver disease leading to more severe hepatic inflammation and fibrosis in chronic hepatitis C which decreases response to IFN therapy.

Ribavarin has also been added as a treatment option with IFN, but ribavirin in thalassemia patients increases transfusion need by a median of 30-40 %, but does not increase major adverse events or treatment withdrawal.

At the end of 2013, the Food and Drug Administration (FDA) approved a new direct-acting antiviral agent for the treatment of HCV infection: Sofosbuvir (Gilead Sciences). Ledipasvir (Gilead Sciences) is a new drug with potent activity against HCV genotypes 1a and 1b. The combination of ledipasvir and sofosbuvir resulted in high rates of response among patients with HCV genotype 1 infection who had received prior treatment with interferon-based regimens. Ledipasvir and sofosbuvir have been combined in a single fixed-dose tablet for use once daily (ledipasvir-sofosbuvir).

Using this drug for HCV therapy alone or in combination with IFN for 12 or 24 weeks, resulted in more than 90% response rates in patients from the general population.

Patients with transfusion-dependent thalassemia major are at increased risk of adverse events with pegylated interferon and ribavirin therapy for HCV due to a notable 30% increase in transfusion requirements during the 48-week therapy. Some patients are not eligible for other treatments as they relapsed or did not respond to previous Ribavarin and IFN regimens. Treatment naïve thalassemia patients with HCV will be exposed to anemia and transfusion-induced iron overload among other adverse events associated with Ribavarin and IFN. These patients in particular, in addition to treatment-naïve thalassemia patients, have limited alternative treatment options available and constitute an area of significant unmet clinical needs. There is currently no literature available showing the efficacy of sofosbuvir/ledipasvir in the treatment of thalassemia patients with hepatitis C. Therefore, this trial will study the efficacy of sofosbuvir/ledipasvir for hepatitis C genotype 1-6 in patients with transfusion-dependent thalassemia.

Ten patients from the Lebanese Chronic Care Center will be enrolled in this open label trial. Patients with transfusion dependent thalassemia with hepatitis C will be enrolled. Study patients will receive the treatment following informed consent and will be followed up regularly by the study coordinator for side effects, compliance and adherence. A blood test for hemoglobin and hematocrit and liver enzyme, will be done on all patients at baseline and then after 4 weeks, 8 weeks , and 12 weeks of therapy. At week 12, levels of the virus in the patient's blood will also be evaluated. Liver imaging will be done throughout the study.

Benefits of this study outweigh potential risks. Side effects of medications used are minor however potential benefits for the patients are possibly treating their hepatitis C with an approved drug (in the general population) at no cost, and for the society, the possibility of finding an oral treatment more efficient and tolerable in this special population.

As for privacy and confidentiality issues, all data will be under lock. The PI and the Co- Investigators will be the only ones with access to that data.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion Dependent thalassemia patients with HCV genotype 1-6
* Age ≥18
* Male and female
* No evidence of hepatocellular carcinoma on ultrasound
* No known drug allergy to the FDA approved drug to be used
* Adequate iron chelation therapy
* Compensated liver disease

Exclusion Criteria:

* Age below 18
* Chronic HCV genotypes 2 or 3
* Allergy to study drug
* Hepatocellular carcinoma
* Inadequate iron chelation therapy
* Decompensated liver disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Response following 12-week therapy (SVR 12) with sofosbuvir/velpatasvir in transfusion-dependent patients with HCV genotype 1-6 | 12 weeks
  Via tests of HepC RNA levels

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No